CLINICAL TRIAL: NCT04530669
Title: The Effect of High Tone Power Therapy on Fatigue and Functional Outcomes in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lama Saad El-Din Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Lama Saad El-Din Mahmoud, Lecturer of physical therapy, Department of Neuromuscular disorders and its surgery, October 6 University
Organization: October 6 University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T. REC/012/002866
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis
Keywords: High Tone Power Therapy; fatigue; functional outcomes
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: active arm and placebo arm; in the active arm patients will receive "high tone power therapy" in addition to the physical therapy conventional selected exercise program, and the placebo arm will receive the same physical exercise program with sham "high tone power therapy".
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): in the active arm patients will receive "high tone power therapy" in addition to the physical therapy conventional selected exercise program
  Interventions: Device: High Tone Power Therapy; Other: exercise program
- control group (Sham Comparator): the sham arm will receive the same physical exercise program with sham "high tone power therapy".
  Interventions: Other: exercise program

INTERVENTIONS:
Device: High Tone Power Therapy — High Tone Power Therapy (HiTop 191): (For group I). The high tone power therapy through using a device (HiTop 191; gbo Medizintechnik, Rimbach, Germany).
  The intensity of the electrical stimulation will be adjusted to a pleasant level that did not produce any pain or discomfort.
  Arms: study group
Other: exercise program — physical therapy conventional selected exercise program inform of functional activities of daily living

SUMMARY:
To investigate the effect of "High Tone Power Therapy" (HTPT) on fatigue and functional outcomes in multiple sclerosis (MS). BACKGROUND: Fatigue and functional limitations considered serious disorders in patients with multiple sclerosis that lead to impairment of the physical activities and disruption of the quality of life (QOL).

HYPOTHESES:

This study hypothesized that:

High Tone Power Therapy will have a significant beneficial effect on fatigue and functional outcomes in in multiple sclerosis

RESEARCH QUESTION:

Is there a beneficial effect of High Tone Power Therapy on fatigue and functional outcomes in multiple sclerosis?

DETAILED DESCRIPTION:
Double blind randomized study including 40 patients with MS. The patients will be randomly allocated into 2 arms: active arm and placebo arm; in the active arm patients will receive "high tone power therapy" in addition to the physical therapy conventional selected exercise program, and the placebo arm will receive the same physical exercise program with sham "high tone power therapy". Either program will be applied 3 times per week for 4 weeks.

The evaluation methods will be done using:

* Expanded Disability Status Scale (EDSS) / Functional Systems Score (FSS),
* Fatigue severity scale and Modified Fatigue Impact Scale. before the exercise program and after finishing the exercise program, The assessor of the patients, before and after the program, will be blinded to the technique used (whether active or sham).

ELIGIBILITY:
Inclusion Criteria:

- Both genders

* Age from 18-50 years
* All MS types will be included (relapsing remitting "RR", secondary progressive "SP, and primary progressive "PP")
* Patients with residual motor / cerebellar / sphincteric impairment that are not responding to conventional pharmacological treatments.
* At least 6 months after the last relapse.
* EDSS from 2-6.5.
* All patients should be receiving a disease modifying therapy with stabilization of the disease course for 1 year in case of SPMS and PPMS.
* Patients that can pay regular visits to the physical center without potential interruption.
* Patients who agree to participate and sign the informed consent. - body mass index (20:29) kg/m2

Exclusion Criteria:

* cognitive impairment that can hinder the ability to communicate or to understand program instructions.
* neurological deficits due to any disease other than MS
* orthopedic abnormalities,
* secondary musculoskeletal complication.
* Patients who refuse participation or signing the informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | 4 weeks
  The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. It is widely used in clinical trials and in the assessment of people with MS.
  The scale was developed by a neurologist called John Kurtzke in 1983 as an advance from his previous 10 step Disability Status Scale (DSS).
  The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist.
  EDSS steps 1.0 to 4.5 refer to people with MS who are able to walk without any aid and is based on measures of impairment in eight functional systems
Functional Systems Score (FSS), | 4 weeks
  On a scale of 0 to 6, the functional system score (FSS) measures how well the major central nervous systems are working and assigns a score to the patient disability. This score uses also information about the gait and use of assistive devices.

CONTACTS AND LOCATIONS:
Overall Officials: Lama S Mahmoud, Study Director — Cairo University; Khalid T Turky, PHD, Study Chair — Ph.D., Assist. prof : Physical Therapy; Nevin M Shalaby, PHD, Study Director — Professor of neurology Department of Neurology , Faculty of Medicine, Cairo University.
Locations (1):
- Kasr Al-Ainy MS clinic, Neurology department, Cairo University hospitals., Al Jīzah, Select State, Egypt

IPD SHARING:
Plan to Share IPD: No